CLINICAL TRIAL: NCT06816342
Title: Assessment of Emergency Spacers Versus Traditional Spacers for Delivery of Aerosolized Drugs
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Omar Ahmed Sayed, Demonstrator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FMBSUREC/01102024/ Hashem
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Asthmatic Patients; MDI; Aerosol Generating Procedure
Keywords: pMDI; valved holding chamber; salbutamol; Aerosol delivery; emergency spacers

STUDY DESIGN:
Intervention Model Description: patients were assigned to 10 groups, each group use a specific type of MDI spacers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- pMDI alone (Active Comparator): patients use pMDI directly without spacer
  Interventions: Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI alone
- Able spacer (Active Comparator): patients use pMDI connected to the Able spacer
  Interventions: Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to Able spacer
- Tips-Haler spacer (Active Comparator): patients use pMDI connected to the Tips-Haler spacer
  Interventions: Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connectec to Tips-Haler spacer
- Aerochaber plus flow vu valved holding chamber (Active Comparator): patients use pMDI connected to the Aerochaber plus flow vu valved holding chamber
  Interventions: Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to Aerochamber plus flow vu valved holding chamber
- Atomizer chamber (Active Comparator): patients use pMDI connected to the Atomizer chamber
  Interventions: Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to Atomizer chamber spacer
- plastic juice cup (Active Comparator): patients use pMDI connected to a plastic juice cup
  Interventions: Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to plastic juice cup spacer
- DispozABLE Spacer (Active Comparator): patients use pMDI connected to the DispozABLE Spacer
  Interventions: Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the DispozABLE spacer
- Lite-Aire Valved holding chamber (Active Comparator): patients use pMDI connected to the Lite-Aire Valved holding chamber
  Interventions: Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the Lite-Aire collapsible valved holding chamber spacer
- ventoline package (Active Comparator): patients use pMDI connected to the ventoline package spacer
  Interventions: Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the MDI package
- paper sheet spacer (Active Comparator): patients use pMDI connected to the paper sheet spacer
  Interventions: Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the hand-made paper sheet spacer

INTERVENTIONS:
Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI alone — patients use ventoline pMDI alone
  Arms: pMDI alone
Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to Able spacer — patients use Ventoline® Evohaler® 100 µg/inhalation pMDI connected to Able spacer
  Arms: Able spacer
Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connectec to Tips-Haler spacer — patients use Ventoline® Evohaler® 100 µg/inhalation pMDI connectec to Tips-Haler spacer
  Arms: Tips-Haler spacer
Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to Aerochamber plus flow vu valved holding chamber — patients use Ventoline® Evohaler® 100 µg/inhalation pMDI connected to Aerochamber plus flow vu valved holding chamber
  Arms: Aerochaber plus flow vu valved holding chamber
Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to Atomizer chamber spacer — patients use Ventoline® Evohaler® 100 µg/inhalation pMDI connected to Atomizer chamber spacer
  Arms: Atomizer chamber
Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to plastic juice cup spacer — patients use Ventoline® Evohaler® 100 µg/inhalation pMDI connected to plastic juice cup spacer
  Arms: plastic juice cup
Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the DispozABLE spacer — patient use Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the DispozABLE spacer
  Arms: DispozABLE Spacer
Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the Lite-Aire collapsible valved holding chamber spacer — patients use Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the Lite-Aire collapsible valved holding chamber spacer
  Arms: Lite-Aire Valved holding chamber
Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the MDI package — patients use Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the MDI package
  Arms: ventoline package
Drug: Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the hand-made paper sheet spacer — patients use Ventoline® Evohaler® 100 µg/inhalation pMDI connected to the hand-made paper sheet spacer
  Arms: paper sheet spacer

SUMMARY:
* The goal of this clinical trial is to evaluate the performance, feasibility, and safety of emergency spacers compared to traditional spacers for the delivery of aerosolized drugs using pMDI. in young children and adult asthmatic patients The main questions it aims to answer are:

  1. Measuring total emitted dose emitted from pMDI alone and attached to spacers.
  2. Determining the pharmacokinetic parameter of aerosol delivered by different spacers.
  3. Determining the lung bioavailability of aerosol delivered by different spacers.
  4. Determining the systemic bioavailability of aerosol delivered by different spacers.
  5. Determining the lung function after aerosol delivered by different spacers.
  6. Determining the safety Researchers will compare salbutamol amount delivered using pMDI alone and pMDI connected to differents spacers to evaluate the performance, feasibility, and safety of emergency spacers compared to traditional spacers for the delivery of aerosolized drugs.

     Participants will asked to
* inhale salbutamol through pMDI alone and pMDI connected to different spacers
* perform lung function test using spirometer
* urine samples will be taken from patients 30 minutes and 24 hours after dose inhalation.
* use pulse oximeter to measure heart rate

DETAILED DESCRIPTION:
I. Introduction Asthma is a chronic inflammatory disease that affects airways and decreases its function. Asthma is the most chronic condition affecting children with increasing prevalence.

Aerosol therapy is the delivery of medication through the inhalation route in the form of fine inhaled particles. Safety is the main advantage of using aerosol, however, there are many limitations related to this route. Among aerosol therapy limitations are low-delivered medication, difficult inhalation techniques of some devices, and patient-related factors. Aerosol-generating devices include nebulizers, dry powder inhalers, and pressurized metered dose inhalers.

Pressurized metered-dose inhalers (pMDIs) are comparatively easy to use and effective. Unfortunately, pMDIs have a significant drawback in that they often lead to inadequate or improper use. pMDI spacers are supplementary devices designed to lessen the issues associated with improper pMDI inhaler technique. By minimizing the need to synchronize inhalation with actuation and enhancing inhaler technique in patients utilizing pMDI, spacers provide an advantage by holding big particles that would typically be deposited in the oropharynx inside the spacer and producing a prolonged aerosol cloud of tiny particles to give the patient more time to inhale following actuation, spacers improve drug targeting. Effective medicine delivery to the airways is especially crucial for elderly and young patients.

The material from which the spacer is made affects the total emitted dose of the inhaled medication. The most popular materials for creating plastic spacers are polypropylene and polycarbonate; however, because they are non-conductive, electrostatic charges are encouraged inside the device. Electrostatic reactions between the electrically charged walls of the spacer and the released medication are inevitable since drugs released from pMDIs are likewise electrically charged. When the charged entities repel each other, the drug particles are forced to go toward the spacer's wall, which lowers the dose that is released.

An essential component that influences the functionality of the spacers is electrostatic charge. The majority of add-on devices on the market are composed of non-conductive material, or "non-antistatic spacers," which gradually build a static charge. Consequently, inventions have been developed to provide antistatic spacers in order to address this issue.

Many traditional forms of spacer are used but with the increased prevalence of asthma, the need for disposable forms of spacers increased. In emergency situations such as exacerbation of pulmonary diseases in busy assembly places as schools and during times of war, any available tool that can be used as disposable spacers would be of important value.

II. Aim of the work This study aims to evaluate the performance, feasibility, and safety of emergency spacers compared to traditional spacers for the delivery of aerosolized drugs using pMDI.

Objectives:

* Measuring total emitted dose emitted from pMDI alone and attached to spacers.
* Measuring the efficacy of different emergency disposable spacer to deliver aerosolized drugs.
* Determining the pharmacokinetic parameter of aerosol delivered by different spacers.
* Determining the lung bioavailability of aerosol delivered by different spacers.
* Determining the systemic bioavailability of aerosol delivered by different spacers.
* Determining the lung function after aerosol delivered by different spacers.
* Measuring heart rate using pulse oximeter to evaluate safety of the amount of salbutamol delivered by different spacers.

III. materials and Methods Type of the study Interventional type IV Site of the study Beni-Suef hospital university - chest diseases department Duration of the study Duration of the study from October 2024 till October 2025 This study will be conducted through 3 models; in-vitro, in-vivo, and ex-vivo models.

The traditional antistatic spacers included the Able valved holding chamber, a 208 mL device manufactured by Clement Clarke International Ltd, UK, designed to optimize drug delivery with minimal static interference. Another antistatic spacer was the Tips-Haler holding chamber, with a capacity of 260 mL, developed by Laboratoire ProtecSom-OptimHal in France, known for its efficiency in maintaining particle integrity. The Aerochamber Plus Flow Vu valved holding chamber, with a volume of 149 mL, produced by Trudell Medical International Europe Ltd, UK, featured a flow indicator to assist in ensuring proper inhalation technique. Additionally, the Atomizer chamber, manufactured by Fox for Medical Engineering, Egypt, represented a non-antistatic option within the traditional category, offering a straightforward design without static mitigation.

The emergency spacers, intended for ad hoc and cost-effective use, included a device constructed from a plastic juice cup, demonstrating the adaptability of readily available materials. The pMDI package, a repurposed Ventolin pMDI casing, offered a practical and accessible solution for immediate use. The Lite-Aire collapsible valved holding chamber, developed by Thayer Medical Corp, provided a portable and disposable option. The DispozABLE paper spacer, created by Clement Clarke International Ltd, UK, was a lightweight and compact alternative suitable for single-use scenarios. Finally, a spacer made from a paper sheet exemplified the simplest form of emergency spacer, leveraging minimal resources for functional delivery support. This diverse selection of devices enabled a comprehensive evaluation of spacer efficacy under varying conditions

* in-vitro model

  1. Total emitted dose The TED was measured using a pMDI sampling apparatus (Copley Scientific Ltd, UK) equipped with a critical flow controller and a 25-mm A/E fiberglass filter (Pall Corporation, USA) within the sampling unit. Inhalation was simulated using a vacuum pump (Brook Crompton, UK) set at a flow rate of 28.3 L·min-¹, replicating breathing volumes of 4 L (adult simulation) and 2 L (older child simulation). Flow rates were controlled using an electronic digital flow meter (MKS Instruments, USA), and all apparatus connections were sealed with Parafilm M (Pechiney Plastic Packaging, USA).

     Before each determination, the pMDI was shaken and primed with two puffs. During testing, the mouthpiece of the pMDI or spacer-pMDI combination was tightly fitted to the sampling unit. For the pMDI alone, drug emission was synchronized with pump activation, while for spacer evaluations, the puff was released into the spacer before activating the pump within 1 second. TED measurements were performed 10 times (n = 10) for each configuration.

     The salbutamol collected on the filter was extracted with 90% acetonitrile and sonicated for 3 minutes, a process validated to recover the full drug dose. Spacers were washed with the same solvent to determine residual drug content. Salbutamol concentrations were quantified using high-performance liquid chromatography (HPLC) with a ZORBAX Eclipse Plus C18 column (Agilent, USA) and a mobile phase of 90:10 acetonitrile-water with 0.1% phosphoric acid, pumped at 1 mL/min. Detection was performed at 225 nm, with calibration ranges from 2 to 100 µg/mL and a lower limit of quantification of 2.5 µg/mL.

     Aerodynamic Particle Size Characterization The aerodynamic particle size of salbutamol was analyzed using the Andersen MKII cascade impactor for the pMDI alone and pMDI-spacer combinations at 4 L and 2 L inhalation volumes. Ten determinations were conducted for each configuration (n = 10). Parameters, including the fine-particle dose (FPD), fine-particle fraction (FPF), and mass median aerodynamic diameter (MMAD), were calculated using CITDAS software (Copley Scientific, UK).
* In-vivo model 120 Mild or moderate asthmatic patients were assigned to 10 groups representing types of spacers used each of 12 patients. A lung function test will be performed before and 15 minutes after dose inhalation for each participant using a spirometer. urine samples 30 minutes after dose inhalation (USAL0.5) and a collective of 24 hours will be taken (USAL24); the first represents lung deposition and the later the systemic bioavailability. USAL0.5 and USAL24 volumes were measured, and aliquots were frozen at -14 °C till treatment and HPLC analysis. Using Oasis mixed-mode cation-exchange (MCX) cartridge (waters Corporation, Milford, Massachusetts), salbutamol was recovered from urine samples via solid-phase extraction. The recovered salbutamol was analyzed by High Performance Liquid Chromatography (HPLC). Heart rate will be measured using a pulse oximeter 15 minutes after dose inhalation to evaluate the safety of the amount of salbutamol delivered.

Inclusion criteria:

* Mild and moderate asthmatic patients aged from 6 - 80 year old.Exclusion criteria:
* Severe asthmatics or patients admitted to an intensive care unit
* ischemic heart disease
* recent abdominal surgery
* inability to perform properly the pulmonary function tests
* hepatic or renal impairment
* hypersensitivity to salbutamol. Sample size technique Sample size is calculated from previous studies using G*Power version 3.1.9.7 (Germany) software.

Sample size calculation:

G*Power software version 3.1.9.7 (Germany) used to detect sample size Using ANOVA: One way test and based on mean and standard deviation of previous published studies with effect size=0.38, α= 0.05, and power=0.8 and found to be 120 participants.

• Ex-vivo model patients are asked to inhale the dose of salbutamol while putting a filter at patients mouth to collect the drug then this filter taken to determine total emitted dose by recovering the drug by centrifugation in 20% acetonitrile then analysed using HPLC.

Statistical analysis Statistical analysis will be done using SPSS program using One way ANOVA test for comparison between different groups.

Ethical consideration: Ethical Approval of the ethical committee at beni-suef university No: FMBSUREC/01102024/ Hashem An informed consent taken from all participants before recruitment in the study, and after explaining the purpose and procedures of the study.

ELIGIBILITY:
Inclusion Criteria:

• Mild and moderate asthmatic patients aged from 6 - 80 year old.

Exclusion Criteria:

* Severe asthmatics or patients admitted to an intensive care unit
* ischemic heart disease
* recent abdominal surgery
* inability to perform properly the pulmonary function tests
* hepatic or renal impairment
* hypersensitivity to salbutamol.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
the total emitted dose | 3 months
  in-vitro determination of the total emitted dose from pMDI alone and different pMDI-spacer combination using pMDI sampling apparatus (Copley Scientific, Nottingham, United Kingdom)
Mass median aerodynamic diameter (MMAD) | 3 months
  in-vitro determination of the aerodynamic particle size of salbutamol after release from the pMDI alone and the pMDI/spacer combinations using Andersen MKII cascade impactor. MMAD will be assessed by CITDAS software (Copley Scientific, Nottingham, UK).
fine particle dose (FPD) | 3 months
  in-vitro determination of the aerodynamic particle size of salbutamol after release from the pMDI alone and the pMDI/spacer combinations using Andersen MKII cascade impactor. fine particle dose (FPD) will be assessed by CITDAS software (Copley Scientific, Nottingham, UK).
fine particle fraction (FPF) | 3 months
  in-vitro determination of the aerodynamic particle size of salbutamol after release from the pMDI alone and the pMDI/spacer combinations using Andersen MKII cascade impactor. fine particle fraction (FPF) will be assessed by CITDAS software (Copley Scientific, Nottingham, UK).
lung bioavailability | 4 months
  lung bioavailability determined by measuring the concentration of salbutamol in urine 30 minutes after dose administration , Salbutamol levels in urine will be measured using HPLC after samples will be solid-phase extracted
systemic bioavailability | 4 months
  systemic bioavailability determined by measuring salbutamol concentration 24 hours collectively after dose administration, Salbutamol levels in urine will be measured using HPLC after samples will be solid-phase extracted

SECONDARY OUTCOMES:
peak expiratory flow (PEF) | 3months
  (PEF) is tested using One flow spirometer before and 15 minutes after dose inhalation.
Forced expiratory volume in second (FEV1) | 3 months
  (FEV1) is tested using One flow spirometer before and 15 minutes after dose inhalation.
forced vital capacity (FVC) | 3 months
  (FVC) is tested using One flow spirometer before and 15 minutes after dose inhalation.
FEV1/FVC ration | 3 months
  FEV1/FVC ration is tested using One flow spirometer before and 15 minutes after dose inhalation.
heart rate | 3 months
  safety determined by measuring heart rate using pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Emam Abdelrahim, professor, Study Chair — Beni-Suef; Haitham Saeed Abdel-Azeez, Associate professor, Study Director — Beni-Suef; Nabila Ibrahim Abdel Mageed Laz, professor, Study Director — Beni-Suef
Locations (1):
- Beni-Suef university hospital, Banī Suwayf, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sayed OA, Laz NI, Abdelrahim ME, Saeed H. Emergency-use spacers: a considerable option for asthmatic patients. Heart Lung. 2026 Jan 2;77:102719. doi: 10.1016/j.hrtlng.2025.102719. Online ahead of print. PMID 41483541